CLINICAL TRIAL: NCT06575777
Title: Analyzing of The Mother And Father's Parenthood Behaviours at The Early Postpartum Period
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Guzin Unlu Suvari, Principal Investigator, Acibadem University
Other Study IDs: 54022451-050.05.04-2019-1810
Record Dates: First submitted 2024-08-27; First posted 2024-08-28 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Parenting; Behavior; Postpartum Period
Keywords: Parenting; Behavior; Postpartum Period
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Married Couples with Newborns: No intervention was applied to the group. The surveys planned to be examined in the postpartum period have been completed.

SUMMARY:
There are many physiological and psychological changes in the postpartum period. One of the changes that occur in the family is the process of becoming a parent. Parenthood is a process that begins with the spouses deciding to get pregnant and continues throughout life. The foundations of an individual's future perspective on themselves and the world are largely determined by the parental interactions they experience in the first year of life and their quality. Parenting behaviors exhibited in the early postpartum period show the extent of communication parents have with their babies in later periods. It is also important because it can have short- and long-term effects on the baby. Parenting behaviors are behaviors in which the mother and father show interest in their baby, such as looking at the newborn baby in the postpartum period, asking questions about the baby, smiling at the newborn baby or making noise. Research shows that these behaviors are affected by socioeconomic reasons, the psychological state of the mother and father, their age, whether the pregnancy was planned, and the general health of the newborn. Parenting behaviors should be observed in the prenatal and postnatal period and supported with education when necessary. Parents need to adapt to their changing roles, develop new relationships, and organize their existing relationships according to their new roles. During the transition to parenthood, in addition to the current home and workplace demands, baby care demands are potential stress factors that can disrupt the organization and process of family life and threaten family and marital functioning. During the parental transition, couples with a greater sense of family cohesion willingly take on the challenges of new parenthood, are committed to seeking meaning in the parenting role, and overcome any challenges encountered during the transition, leading to a more satisfying family and marital relationship. Additionally, spousal support and involvement in infant care have been found to be associated with higher satisfaction in marital relationships and family functioning. Research suggests that spousal involvement and support for each other are particularly important for family and marital functioning during the transition to parenthood. Although significant research has been conducted on family and marital functioning during the transition to the parenting role, research on the effects of family cohesion, social support, and stress during the perinatal period on family and marital functioning is limited. This study aimed to examine the parenting behaviors and marital adjustment of mothers and fathers during the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Having a full-term birth (38-42 weeks of gestation)
* No high-risk pregnancy
* Having a healthy newborn
* The couple being married

Exclusion Criteria:

* Illiteracy
* High-risk pregnancy
* Multiple pregnancy
* Prematurity
* Newborn weighing less than 2500g or more than 4000g

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The research population consisted of married couples who had recently given birth.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Sociodemographic and Obstetric Data Collection Form for Mothers | Baseline (completed at the first meeting with the mother, either before birth in planned births or on Day 1 after birth in unplanned births).
  This form, prepared by the researcher through a literature review, consists of 18 questions and is designed to obtain sociodemographic and obstetric information from the mothers participating in the study.
Sociodemographic and Obstetric Data Collection Form for Fathers | Baseline (completed at the first meeting with the father, either before birth in planned births or on Day 1 after birth in unplanned births).
  This form, prepared by the researcher through a literature review, consists of 9 questions and is designed to obtain sociodemographic information from the fathers participating in the study.
Marital Adjustment Scale | Baseline (completed at the first meeting with the participant, either before birth in planned births or on Day 1 after birth in unplanned births).
  The Marital Adjustment Scale consists of 15 items and is used to assess marital adjustment. The scale yields a total score ranging from 1 to 60, with scores of 43 and above indicating marital adjustment and scores below 43 indicating marital maladjustment.
Postpartum Parenting Behavior Scale | Day 1 (assessed during the first 10 minutes of the parent and newborn's first encounter).
  The Postpartum Parenting Behavior Scale is used to assess parenting behaviors during the first encounter between parents and their newborn. The scale measures behaviors like close contact, affectionate touch, and positive comments through a 10-minute observation, with each item scored as present or absent. The total score ranges from 0 to 6, with higher scores indicating more positive parenting behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Selinay Aktaş Demir, Ph. D. (C), Principal Investigator — İstinye University; Anayit Margirit Coşkun, Prof. Dr., Principal Investigator — İstanbul Atlas University; Dilek Sinem Uludağ, B.Sc. (Midwife), Principal Investigator — Esenler Maternity and Children's Hospital
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared online via Mendeley Data when requested from the responsible researcher by email.
URL: https://data.mendeley.com/

REFERENCES:
- [Background] Claridge, A. M., Lettenberger-Klein, C. G., & VanDonge, C. M. (2017). Pregnancy intention and positive parenting behaviors among first-time mothers: The importance of mothers' contexts. Journal of Family Issues, 38(7), 883-903.
- [Background] Aslan, E., Erturk, S., Demir, H., & Aksoy, O. (2017). Fathers' attachment status to their infants. International Journal of Caring Sciences, 10(3), 1410-1418.
- [Background] Avcı, S. Ç., & Cetişli, N. E. (2021). Effect of birth type on parenting behavior, infant perception and maternal attachment. Cukurova Medical Journal, 46(3), 1059-1069.
- [Background] Bilgin, Z., & Alpar, Ş. E. (2018). Kadınların maternal bağlanma algısı ve anneliğe ilişkin görüşleri/The relationship between maternal attachment perception of women's maternal role. Sağlık Bilimleri ve Meslekleri Dergisi, 5(1), 6-15.
- [Background] Çalışır, H., Karaçam, Z., Akgül, F. A., & Kurnaz, D. A. (2009). Doğum sonrası ebeveynlik davranışı ölçeği'nin türkçe formunun geçerliği ve güvenirliği. Journal of Anatolia Nursing and Health Sciences, 12(1).
- [Background] Endendijk JJ, Groeneveld MG, Bakermans-Kranenburg MJ, Mesman J. Gender-Differentiated Parenting Revisited: Meta-Analysis Reveals Very Few Differences in Parental Control of Boys and Girls. PLoS One. 2016 Jul 14;11(7):e0159193. doi: 10.1371/journal.pone.0159193. eCollection 2016. PMID 27416099
- [Background] Ergin A, Özdilek R. (2014). Değişen babalık rolü ve erkek sağlığına etkileri. Hemşirelikte Eğitim ve Araştırma Dergisi. 11:3-8.
- [Background] Güneş, E., & Işık, C. (2023). Maternal-paternal bağlanmayı etkileyen faktörler ve ebelik yaklaşımları. Sağlık Profesyonelleri Araştırma Dergisi, 5(1), 89-95.
- [Background] Kaur, T., & Bhargava, M. (2016). Correlates of marital harmony. Indian Journal of Health and Wellbeing, 7(9), 893.
- [Background] Kaya, A. G., & Buğa, A. (2021). Anne babaların ebeveyn davranışlarının ve evlilik doyumlarının incelenmesi. Sosyal Politika Çalışmaları Dergisi, 21(51), 371-410.
- [Background] Kaya, C. E., & Şahin, N. H. (2020). Ebeveyn uyum desteği programı ile ebeveyn öz yeterlik algısının geliştirilmesi. Ordu Üniversitesi Hemşirelik Çalışmaları Dergisi, 3(3), 319-328.
- [Background] Kışlak, T. Ş. (1999). Evlilikte Uyum Ölçeğinin (EUÖ) güvenirlik ve geçerlik çalışması. Psikiyatri Psikoloji Psikofarmakoloji Dergisi, 7(1), 50-57.
- [Background] Lazoğlu, M., Gümüşdaş, M., & Apay, S. E. (2022). X, Y, Z Kuşağı Lohusaların Ebeveynlik Davranışlarının Karşılaştırılması. Jinekoloji-Obstetrik ve Neonatoloji Tıp Dergisi, 19(1), 1169-1175.
- [Background] Koç, Ö., Özkan, H., & Bekmezci, H. (2016). Evaluating the correlation between maternal role and parenting behavior. İzmir Dr. Behçet Uz Çocuk Hast. Dergisi 2016; 6(2):143-150.
- [Background] Locke, H. J., & Wallace, K. M. (1959). Short marital-adjustment and prediction tests: Their reliability and validity. Marriage and Family Living, 21(3), 251-255.
- [Background] Menendez S, Hidalgo MV, Jimenez L, Moreno MC. Father involvement and marital relationship during transition to parenthood: differences between dual and single-earner families. Span J Psychol. 2011 Nov;14(2):639-47. doi: 10.5209/rev_sjop.2011.v14.n2.12. PMID 22059310
- [Background] Mutlu B, Erkut Z, Yildirim Z, Gundogdu N. A review on the relationship between marital adjustment and maternal attachment. Rev Assoc Med Bras (1992). 2018 Mar;64(3):243-252. doi: 10.1590/1806-9282.64.03.243. PMID 29641776
- [Background] Nelson JA, O'Brien M. Does an Unplanned Pregnancy have Long-Term Implications for Mother-Child Relationships? J Fam Issues. 2012 Apr;33(4):506-526. doi: 10.1177/0192513X11420820. Epub 2011 Sep 1. PMID 28179747
- [Background] Özdemir, A. A., Köse, S., Küçükoğlu, S., & Akbakay, S. (2021). Türkiye'nin Doğusunda Bir İlde Yaşayan Annelerin Doğum Sonu Dönemde Ebeveynlik Davranışları. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 24(2), 231-238
- [Background] Özkan, H., Çelebioğlu, A., Üst, Z. D., & Kurudirek, F. (2016). Doğum sonu dönemde babaların ebeveynlik davranışlarının incelenmesi. İzmir Dr. Behçet Uz Çocuk Hast. Dergisi, 6(3), 191-196.
- [Background] Planalp EM, Van Hulle CA, Goldsmith HH. Parenting in context: Marital adjustment, parent affect, and child temperament in complex families. J Fam Psychol. 2019 Aug;33(5):532-541. doi: 10.1037/fam0000511. Epub 2019 Feb 7. PMID 30730182
- [Background] Salmela-Aro K., Nurmi J.-E., Saisto T. & Halmesmäki E. (2010) Spousal support for personal goals and relationship satisfaction among women during the transition to parenthood. International Journal of Behavioral Development 34, 229-237.
- [Background] Schaber R, Kopp M, Zahringer A, Mack JT, Kress V, Garthus-Niegel S. Paternal Leave and Father-Infant Bonding: Findings From the Population-Based Cohort Study DREAM. Front Psychol. 2021 Jun 4;12:668028. doi: 10.3389/fpsyg.2021.668028. eCollection 2021. PMID 34149562
- [Background] Yu CY, Hung CH, Chan TF, Yeh CH, Lai CY. Prenatal predictors for father-infant attachment after childbirth. J Clin Nurs. 2012 Jun;21(11-12):1577-83. doi: 10.1111/j.1365-2702.2011.04003.x. Epub 2012 Mar 12. PMID 22409833